CLINICAL TRIAL: NCT05644106
Title: Listening Benefits From a Hearing-aid App, a Personal Sound Amplification Product, and a Hearing Aid in Hearing-impaired Listeners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Moo Kyun, Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2105-200-1223
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hearing Disorders
Keywords: Hearing aid, Personal sound amplification product, Hearing aid application, Hearing loss
MeSH Terms: conditions — Hearing Disorders; Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unaided (Active Comparator)
  Interventions: Device: personal sound amplification product, hearing aid
- Aided (Active Comparator)
  Interventions: Device: personal sound amplification product, hearing aid

INTERVENTIONS:
Device: personal sound amplification product, hearing aid — the device for hearing gain in sensorineural hearing loss

SUMMARY:
Interest and demand for sound amplifiers are increasing due to the burden of purchasing hearing aids and technological advances in healthcare products, and the demand is expected to increase rapidly. For sensorineural hearing loss patients, who are subject to wearing hearing aids, it aims to compare the effect of hearing aid application and personal sound amplification product (PSAPs) compared to the hearing aids

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 20 who speak Korean as their mother tongue and have no mental or physical limitations in conducting test.
2. Hearing loss patients with a hearing threshold of 26 dB or higher in the four frequency (0.5, 1, 2, 4 kHz)
3. Those who do not have a history of neurological disease, cognitive disorder, learning disorder, or language disorder at the time of recruitment

Exclusion Criteria:

1. In case that communication is difficult, equipment cannot be handled, or it is difficult to cooperate with the inspection
2. Acoustic nerve lesions or central nervous system disease
3. Those suspected of having false hearing loss
4. Those who have secondary benefits related to clinical trials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2023-08-09 (Estimated)

PRIMARY OUTCOMES:
The hearing level threshold (decibel) after each treatment | 1 month
  The comparison of hearing threshold, which is calculated as mean decibel on four frequencies, among different treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jo S, Park MK, Seo JH, Lee KE, Han JS, Lim JH, Lee JH, Oh SH. Feasibility of a Smartphone-Based Hearing Aid App for Mild-to-Moderate Hearing Loss: Prospective Multicenter Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Oct 5;11:e46911. doi: 10.2196/46911. PMID 37800887